CLINICAL TRIAL: NCT05605379
Title: CML Pediatric ITK Response According to Molecular Identification at Diagnosis (CML Piramid
Brief Title: CML Pediatric ITK Response According to Molecular Identification at Diagnosis
Acronym: CML Piramid
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2022/44
Record Dates: First submitted 2022-10-12; First posted 2022-11-04 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Chronic Myeloid Leukemia; Children; Molecular landscape; TKI response; Expression profile
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — High-Throughput Nucleotide Sequencing; DNA; RNA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Responders (with CCR at 1 year)
  Interventions: Biological: Next Generation Sequencing (DNA and RNA)
- No responders (without CCR at 1 year)
  Interventions: Biological: Next Generation Sequencing (DNA and RNA)

INTERVENTIONS:
Biological: Next Generation Sequencing (DNA and RNA) — Targeted Next Generation Sequencing (DNA and RNA)

SUMMARY:
Treatment of chronic myeloid leukemia (CML) has been revolutionized by tyrosine kinase inhibitor (TKI). Nevertheless, case of failure and suboptimal response are still observed even in children. Pediatric CML is a rare disease and differs from adult in terms of disease presentation and treatment response underlying a likely different CML biology. Molecular mechanisms that induce resistance to TKI are still poorly characterized except mutations in the tyrosine kinase domain of BCR::ABL1. We propose to search for a molecular signature to predict the response to TKI in the pediatric population.

DETAILED DESCRIPTION:
Commonly mutated genes associated with myeloid malignancies have been described in acceleration phase and blastic phase but also at diagnostic in adult chronic phase-CML (CP-CML). The impact of these mutations on treatment response is still debated but several studies observed a worse outcome in adult patients with some mutations. In children only one study explored the molecular status of 30 genes in 21 children and young adults. They found a higher proportion of ASXL1 mutations in children than in adult They did not observed any significant difference in overall survival of ASXL1 mutated versus non-mutated patients but probably due the small size of the cohort. We propose here, to investigate retrospectively on DNA at diagnosis of 88 CP-CML children the mutation status of 64 genes by next generation sequencing and to see if there is an association with the response to TKI treatment. We will complete the molecular signature by analyzing the differentially genetic expression profile by RNA-seq on peripheral blood RNA of 8 patients with CCR at 12 months (and/or a BCR ::ABL1 IS ≤1%IS) and 8 patients with no CCR at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age at diagnosis less than or equal to 18 years
* Presence of a Philadelphia chromosome detected by cytogenetic analysis (conventional karyotype or Fluorescence In Situ Hybridization (FISH)) and a BCR ::ABL1 transcript e13a2 ou e14a2
* Diagnosis in chronic phase according to the European Leukemia Net (ELN) criteria
* First-line treatment with TKIs
* Possible pre-treatment with hydroxyurea
* DNA available at diagnosis
* RNA available for a sub-group patients (8 responders vs 8 no responders)

Exclusion Criteria:

* Age at diagnosis more than 18 years
* Diagnosis in accelerated phase or blastic phase
* First line treatment other than TKI

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric CML patients
Sampling Method: Non-Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Complete cytogenetic response (CCR) | At 12 months from TKI start
  We will analyse the impact of the presence of mutations on the obtention of CCR

SECONDARY OUTCOMES:
Molecular response | At 3, 12, 18 and 24 months
  We will analyse the impact of the presence of mutations on the obtention of molecular response (MR4, MMR)
Type of response according to ELN2020 criteria | At 3, 12, 18 and 24 months
  We will analyse the impact of the presence of mutations on the type of response
Occurrence of secondary resistance | At 3, 12, 18 and 24 months
  We will analyse the impact of the presence of mutations on the occurrence of loss of complete hematologic, and/or cytogenetic and/or molecular responses
Occurrence of TK domain mutation | At 3, 12 18 and 24 months
  We will analyse the impact of the presence of mutations on the occurrence of mutation in the TK domain ABL1
Progression Free Survival (PFS) | At 3, 12, 18 and 24 months
  Progression to accelerated phase or blast crisis and deaths will be analysis according to the mutational status
Overall Survival (OS) | At 3, 12, 18 and 24 months
  We will analyse the impact of the presence of mutations on OS

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Service Hématologie Biologique, Bordeaux, France